CLINICAL TRIAL: NCT01003977
Title: REWARDS (Registry Experience at the Washington Hospital Center, DES - Xience V)
Brief Title: Registry Experience at the Washington Hospital Center, DES - Xience V
Acronym: REWARDS XV
Status: Completed | Type: Observational
Sponsor: Rebecca Torguson (Other)
Responsible Party: Sponsor-Investigator, Rebecca Torguson, Director, ACRO, Medstar Health Research Institute
Organization: Medstar Health Research Institute (Other)
Other Study IDs: REWARDS XV
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xience V: Patients treated with a Xience V everolimus-eluting stent

SUMMARY:
Single center registry of patients who have received a Xience V everolimus-eluting stent at the Washington Hospital Center, with the primary objective to assess clinical success and safety at 30 days, 6 months and 1 year post-implantation.

DETAILED DESCRIPTION:
Interventional cardiology was revolutionized by the invention of stents, initially with the bare-metal stents (BMS) and recently with the drug-eluting stents (DES). The everolimus eluting, Xience V stents have shown very promising results in randomized clinical trials, demonstrating a reduction of clinical and angiographic restenosis in comparison to BMS, and comparable clinically-driven target lesion revascularization rates in comparison with sirolimus-eluting stents. While registry data is available from outside of the United States, it will be important to collect "real-world" data regarding the stent usage and outcomes in the United States. In this study we propose to follow patients who received at least one Xience V® Stent for at least 1 year post initial stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, >18 years of age
* Patients who received at least one Xience V drug-eluting stent at the Washington Hospital Center

Exclusion Criteria:

* Patients who received another type of DES (other than Xience V) or a bare metal stent at the time of initial Xience V stent implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a Xience V, everolimus-eluting, Stent at the Washington Hospital Center.
Sampling Method: Non-Probability Sample
Enrollment: 6069 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of Major Adverse Cardiac Events (MACE) post Xience V implantation | Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Research Institute/Cardiovascular Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States